CLINICAL TRIAL: NCT01030419
Title: Activity, Gait, and Efficacy (AGE II): Functional Limitations and Quality of Life
Acronym: AGE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Edward McAuley, Professor, Kinesiology and Community Health, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UIUC_IRB_09765; 2R01AG020118-05A2 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Aging
Keywords: Aging; Quality of Life; Functional fitness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FlexToBa physical activity DVD (Experimental): Participants in this arm will receive a physical activity program delivered by DVD that focuses on exercises targeting flexibility, toning and balance. These exercises will be progressive in nature throughout the six months and will also focus on modifications for all ability levels. Participants will be provided with three DVDs including: an Introduction to physical activity, Sessions 1-3, and Sessions 4-6, which they will be asked to watch and participate in over the course of six months.
  Interventions: Behavioral: Home-based, DVD-delivered physical activity
- Usual care-Wait list (Placebo Comparator): Participants in this arm will receive a DVD that focuses on healthy aging topics but does not include physical activity. They will receive the FlexToBa DVD after the completion of the 12-month follow-up testing.
  Interventions: Behavioral: Usual care/Wait list

INTERVENTIONS:
Behavioral: Home-based, DVD-delivered physical activity — Subjects will be participating in a home-based physical activity program that focuses on flexibility, toning and balance. Exercises will be progressive over the six-months and will highlight modifications for varying levels. This program will be delivered on 3 DVDs. Participants will be asked to exercise with the DVD at least three times per week. Additionally, they will be encouraged to add two days of aerobic activity (e.g. walking) each week.
  Arms: FlexToBa physical activity DVD
Behavioral: Usual care/Wait list — Participants in this arm will receive a DVD that focuses on healthy aging topics but does not include physical activity. They will receive the FlexToBa DVD afer the completion of the 12-month follow-up testing.
  Arms: Usual care-Wait list

SUMMARY:
The purpose of this study is to test the effectiveness of a DVD-delivered, home-based, six-month physical activity intervention for older adults.

A comparative effectiveness study of the FlexToBa DVD exercise program will be conducted in 2014.

DETAILED DESCRIPTION:
This program compares progressive strength, flexibility, toning and balance (FlexToBa) activities delivered via home-based DVD intervention compared to an attention control group to determine the program's effects on functional limitations, functional performance in everyday activities, balance, and quality of life (QOL) in sedentary older adults over 65 years of age. The principals of REAIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) will be implemented into the design and evaluation of the program in order to determine the generalizable cost-effectiveness and potential public health impact of delivering physical activity to older adults via DVD media. Measurements assessed at baseline, six months, and 12 months include: functional performance and functional limitations, self-efficacy, physical activity, and measures of health status and well-being. We propose to recruit and randomly assign 250 older (65+) adults from across Central Illinois to the FlexToBa condition or to an attention control condition. The former will receive the activity program DVD and the latter will receive a healthy aging DVD (with no physical activity instruction). The control group will be offered the FlexToBa program following 6-month follow-up assessments. The health relevance of this project is considerable as it targets a population that is largely sedentary and suffers from unprecedented levels of functional limitations, factors that have significant implications for compromised quality of life and independent living. By adopting broad recruitment strategies with few exclusionary criteria, we will be able to effectively improve the physical activity behavior of a diverse class of older adults. Offering this as a DVD-based physical activity program will provide a convenient opportunity for older adults to become and stay physically active. We intend to provide a limited number of DVD players to those interested participants who do not already own one.

In 2014, investigators will study the comparative effectiveness of the FlexToBa DVD trial as compared to a DVD-only intervention.Researchers will provide the exercise DVD to an entire wave/group of participants with half receiving the motivational telephone calls and feedback (as with earlier waves) and the other half receiving no motivational communications.

The procedures for the Support Group, who receive the motivational support, will be identical to earlier waves. Both groups will receive the FlexToBa DVDs and equipment at the initial testing and orientation meeting but the Effectiveness Group will not receive the motivational feedback. Testing at month six is identical to earlier waves and both groups will be asked to evaluate the program at the end of the intervention.

There is no plan for follow-up testing at month 12 or month 24 for this wave of participants.

ELIGIBILITY:
Inclusion Criteria:

* being non-active, defined as reporting not engaging in regular activity (30 minutes accumulated per day) on more than two days of the week in the prior six months;
* aged 65 - 85 years;
* capable of participation in a program of flexibility,
* toning and balance without exacerbating any pre-existing conditions;
* able to obtain medical clearance for physical activity.

Exclusion Criteria:

* self-reported physical activity on a regular basis within the last six months (2 times or more per week);
* any physical disability that strictly prohibits stretching, strengthening and balance exercises;
* no regular access to a television;
* unable to successfully answer 21 out of 39 questions on the Telephone Interview of Cognitive Status questionnaire (TICS-M).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 410 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Functional performance, balance and reduced self-reported upper and lower body functional limitations in sedentary, older adults' physical activity. | Baseline, 6-month, 12-month follow-up

SECONDARY OUTCOMES:
Quality of Life | Baseline, 6-month, 12-month follow-up
Self-efficacy | Baseline, six-months, and 12-month folluw-up
REAIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) to determine the impact of delivering physical activity via DVD media | Baseline, 6-months, 12-month follow-up
Adherence | Baseline, 6-months, 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salerno EA, Gothe NP, Fanning J, Peterson LL, Colditz GA, McAuley E. Effects of a DVD-delivered randomized controlled physical activity intervention on functional health in cancer survivors. BMC Cancer. 2021 Jul 29;21(1):870. doi: 10.1186/s12885-021-08608-8. PMID 34325676
- [Derived] Aguinaga S, Ehlers DK, Salerno EA, Fanning J, Motl RW, McAuley E. Home-Based Physical Activity Program Improves Depression and Anxiety in Older Adults. J Phys Act Health. 2018 Sep 1;15(9):692-696. doi: 10.1123/jpah.2017-0390. Epub 2018 Apr 6. PMID 29625012
- [Derived] Awick EA, Ehlers D, Fanning J, Phillips SM, Wojcicki T, Mackenzie MJ, Motl R, McAuley E. Effects of a Home-Based DVD-Delivered Physical Activity Program on Self-Esteem in Older Adults: Results From a Randomized Controlled Trial. Psychosom Med. 2017 Jan;79(1):71-80. doi: 10.1097/PSY.0000000000000358. PMID 27359182
- [Derived] Roberts S, Awick E, Fanning JT, Ehlers D, Motl RW, McAuley E. Long-Term Maintenance of Physical Function in Older Adults Following a DVD-Delivered Exercise Intervention. J Aging Phys Act. 2017 Jan;25(1):27-31. doi: 10.1123/japa.2015-0284. Epub 2016 Aug 24. PMID 27180818
- [Derived] Fanning J, Awick EA, Wojcicki TR, Gothe N, Roberts S, Ehlers DK, Motl RW, McAuley E. Effects of a DVD-Delivered Exercise Intervention on Maintenance of Physical Activity in Older Adults. J Phys Act Health. 2016 Jun;13(6):594-8. doi: 10.1123/jpah.2015-0173. Epub 2015 Nov 23. PMID 26595937
- [Derived] McAuley E, Wojcicki TR, White SM, Mailey EL, Szabo AN, Gothe N, Olson EA, Mullen SP, Fanning J, Motl RW, Rosengren K, Estabrooks P. Physical activity, function, and quality of life: design and methods of the FlexToBa trial. Contemp Clin Trials. 2012 Jan;33(1):228-36. doi: 10.1016/j.cct.2011.10.002. Epub 2011 Oct 17. PMID 22024470